CLINICAL TRIAL: NCT05909579
Title: Investigating the Effectiveness of PelvicSense(R) on Pain and Sexual Outcomes in Endometriosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Caroline Pukall (Other)
Responsible Party: Sponsor-Investigator, Dr. Caroline Pukall, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 379631-2
Record Dates: First submitted 2023-05-05; First posted 2023-06-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3 month PelvicSense(R) program (Experimental): PelvicSense® is a home-based physiotherapy program integrating multiple techniques, including relaxation, breathing, stretching, strengthening and at-home manual therapy. This program also educates participants about the anatomy and physiology of the pelvis and teaches strategies to strengthen the mind-muscle connection to the pelvis.
  Interventions: Behavioral: PelvicSense (R)

INTERVENTIONS:
Behavioral: PelvicSense (R) — PelvicSense® is a home-based physiotherapy program integrating multiple techniques, including relaxation, breathing, stretching, strengthening and at-home manual therapy. This program also educates participants about the anatomy and physiology of the pelvis and teaches strategies to strengthen the mind-muscle connection to the pelvis.

SUMMARY:
This study will examine the effectiveness of the PelvicSense 3-month online program on pain and other outcomes in those with endometriosis. This study is prospective in nature and will involve several assessment points: baseline, immediately post-treatment (at the end of the 3 month program), and 3-month follow up. All aspects of the study will be conducted remotely (e.g., online, email, video calls), and participants will be at least 18 years of age, fluent in English, and experience pain due to endometriosis for at least 3 months with a physician diagnosis. Participants are expected to continue their treatment as usual and this information will be documented throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, fluent in English, and have a formal diagnosis of endometriosis for at least 3 months.

Exclusion Criteria:

* Younger than 18 years of age, nonfluency in English, self-identified diagnosis, endometriosis duration of less than 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All identities accepted with female pelvic anatomy.
Enrollment: 50 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Pain Intensity Numerical Rating Scale (NRS). Participants will be asked to report their pain intensity on an 11-point numerical scale of 0 (no pain) to 10 (worst pain ever felt).
Pain intensity | At the end of the 3 month program
  Pain Intensity Numerical Rating Scale (NRS). Participants will be asked to report their pain intensity on an 11-point numerical scale of 0 (no pain) to 10 (worst pain ever felt).
Pain intensity | 3 months after the end of the program
  Pain Intensity Numerical Rating Scale (NRS). Participants will be asked to report their pain intensity on an 11-point numerical scale of 0 (no pain) to 10 (worst pain ever felt).

SECONDARY OUTCOMES:
Pain catastrophizing | Baseline
  Pain Catastrophizing Scale (PCS). 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.
Pain catastrophizing | At the end of the 3 month program
  Pain Catastrophizing Scale (PCS). 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.
Pain catastrophizing | 3 months after the end of the program
  Pain Catastrophizing Scale (PCS). 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.

OTHER OUTCOMES:
Sexual distress | Baseline
  Sexual Distress Scale, Short Form (SDS-SF). 5 items rated on 5 point scales from 0 (never) to 4 (always). Total scores range from 0-20. Higher scores are worse.
Sexual distress | At the end of the 3 month program
  Sexual Distress Scale, Short Form (SDS-SF). 5 items rated on 5 point scales from 0 (never) to 4 (always). Total scores range from 0-20. Higher scores are worse.
Sexual distress | 3 months after the end of the program
  Sexual Distress Scale, Short Form (SDS-SF). 5 items rated on 5 point scales from 0 (never) to 4 (always). Total scores range from 0-20. Higher scores are worse.
Pain self-efficacy | Baseline
  Pain Self-Efficacy Questionnaire (PSEQ). 10 items rated on 7 point scales from 0 (not at all confident) to 6 (completely confident). Total scores range from 0-60.
Pain self-efficacy | At the end of the 3 month program
  Pain Self-Efficacy Questionnaire (PSEQ). 10 items rated on 7 point scales from 0 (not at all confident) to 6 (completely confident). Total scores range from 0-60.
Pain self-efficacy | 3 months after the end of the program
  Pain Self-Efficacy Questionnaire (PSEQ). 10 items rated on 7 point scales from 0 (not at all confident) to 6 (completely confident). Total scores range from 0-60.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Pukall, PhD, Principal Investigator — Queen's University
Locations (1):
- Sexual Health Research Laboratory, Department of Psychology, Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to other researchers after publication of the results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be available to other researchers for 2 years after publication of the results.
Access Criteria: Please email the PI at caroline.pukall@queensu.ca